CLINICAL TRIAL: NCT03302078
Title: Relative Bioavailability of BI 1015550 Following Oral Administration Under Fed and Fasted Conditions in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0020; 2017-002271-26 (EudraCT Number)
Record Dates: First submitted 2017-09-28; First posted 2017-10-04 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 1015550 24 milligrams (mg) fed / BI 1015550 24 mg fast (Experimental): Subjects were treated orally in period 1 with single dose of BI 1015550 4x6 mg (24 mg) tablets under fed condition, followed in period 2 with 4x6 mg (24 mg) of BI 1015550 tablets under fasted condition, each treatment with 240 milliliter (mL) water, separated by a wash-out period of at least 7 days between drug administrations.
  Interventions: Drug: BI 1015550
- BI 1015550 24 mg fast / BI 1015550 24 mg fed (Experimental): Subjects were treated orally in period 1 with single dose of BI 1015550 4x6 mg (24 mg) tablets under fasted condition, followed in period 2 with 4x6 mg (24 mg) of BI 1015550 tablets under fed condition, each treatment with 240 mL water, separated by a wash-out period of at least 7 days between drug administrations.
  Interventions: Drug: BI 1015550

INTERVENTIONS:
Drug: BI 1015550 — Single dose of BI 1015550 4x6 mg (24 mg) tablets under fed or fasted condition
  Other Names: Nerandomilast; JASCAYD®

SUMMARY:
The primary objective of this trial is to investigate the effect of food on the pharmacokinetics of the oral tablet formulation of BI 1015550 by investigating the relative bioavailability of TF1 under fed and fasted conditions.

The assessment of safety and tolerability will be an additional objective of this part.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders including but not limited to mood disorders and any signs of suicidality (ideation as well as behavior) in the past
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant Electrocardiogram (ECG) finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects who do not agree to minimize the risk of female partners becoming pregnant from the first dosing day until two month after the study completion. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device, hormonal contraceptive since at least two month)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-12-13 (Actual); Study Completion 2017-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases(in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a phase I, open-label, randomised, single dose, two-period, two-sequence crossover trial performed in healthy subjects.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial. Participants attended specialist site which would then ensure that all participants met all inclusion/exclusion criteria. Participants were not to be entered to trial treatment if any one of the specific entry criteria were not met
Period: Treatment Period 1
Arm/Group | BI 1015550 24 milligrams (mg) fed / BI 1015550 24 mg fast | BI 1015550 24 mg fast / BI 1015550 24 mg fed
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | BI 1015550 24 milligrams (mg) fed / BI 1015550 24 mg fast | BI 1015550 24 mg fast / BI 1015550 24 mg fed
Started | 6 | 6
Completed | 6 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Treatment Period 2
Arm/Group | BI 1015550 24 milligrams (mg) fed / BI 1015550 24 mg fast | BI 1015550 24 mg fast / BI 1015550 24 mg fed
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were randomised and treated with at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 1015550 24 Milligrams (mg) Fed / BI 1015550 24 mg Fast | BI 1015550 24 mg Fast / BI 1015550 24 mg Fed | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (8.1) | 40.5 (13.1) | 43.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 to the last quantifiable data point. Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequence', 'period', and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Adjusted mean estimates and their difference on log-scale were back-transformed to the original scale.
Time Frame: Pharmacokinetic samples were collected at 3:00 (hours:minutes) before and 0:15, 0:30, 0:45, 1:00, 1:15, 1:30, 2:00, 3:00, 4:00, 6:00, 8:00, 12:00, 24:00, 34:00, 48:00, 72:00, 96:00 and 120:00 (hours:minutes) after drug administration on day 1.
Population: Pharmacokinetic (PK) set (PKS):The PKS included all subjects in the Treated Set (TS) who provided at least one primary or secondary PK parameter that was not excluded due to important protocol violations relevant to the evaluation of PK or due to PK non-evaluability.
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole*hours/Liter (nmol*h/L)
Groups:
- BI 1015550 24 mg fed (Test, T): Subjects were treated orally with single dose of BI 1015550 4x6 milligrams (mg) (24 mg) tablets with 240 mL of water under fed condition on day 1.
- BI 1015550 24 mg fast (Reference, R): Subjects were treated orally with single dose of BI 1015550 4x6 mg (24 mg) tablets with 240 mL of water under fast condition on day 1.
Arm/Group | BI 1015550 24 mg fed (Test, T) | BI 1015550 24 mg fast (Reference, R)
Number analyzed (Participants) | 11 | 12
nanomole*hours/Liter (nmol*h/L) | 4164.32 (NA) — Adjusted geometric standard error = 1.06 | 4057.42 (NA) — Adjusted geometric standard error = 1.06
Statistical Analysis 1: Comparison: BI 1015550 24 mg fed (Test, T) vs BI 1015550 24 mg fast (Reference, R); The analysis of variance (ANOVA) model on a logarithmic scale included effects accounting for the following sources of variation: 'sequence', 'subjects within sequence', 'period', and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. No hypothesis was tested and no acceptance range was specified. This was an intra-individual assessment and actually only 12 subjects were analyzed; Test type: Other; Geometric Mean (T/R) ratio (%) = 102.63, 90% CI 2-sided [98.31 to 107.15] — To get geometric mean ratio and confidence interval, least square estimates of log-transformed PK endpoint for T and R were back transformed to original scale. Intra-individual geometric coefficient of variance (%) = 5.5

2. Primary Outcome: Maximum Measured Concentration of BI 1015550 in Plasma (Cmax)
Description: Cmax, maximum measured concentration of BI 1015550 in plasma. Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequence', 'period', and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Adjusted mean estimates and their difference on log-scale were back-transformed to the original scale.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomole/Liter (nmol/L)
Arm/Group | BI 1015550 24 mg fed (Test, T) | BI 1015550 24 mg fast (Reference, R)
Number analyzed (Participants) | 11 | 12
nanomole/Liter (nmol/L) | 404.34 (NA) — Adjusted geometric standard error = 1.06 | 511.29 (NA) — Adjusted geometric standard error = 1.06
Statistical Analysis 1: Comparison: BI 1015550 24 mg fed (Test, T) vs BI 1015550 24 mg fast (Reference, R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean (T/R) ratio (%) = 79.08, 90% CI 2-sided [69.96 to 89.40] — To get geometric mean ratio and confidence interval, least square estimates of log-transformed PK endpoint for T and R were back transformed to original scale. Intra-individual geometric coefficient of variance (%) = 16.0

3. Secondary Outcome: Area Under the Concentration-time Curve of BI 1015550 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: AUC0-inf, area under the concentration-time curve of BI 1015550 in plasma over the time interval from 0 extrapolated to infinity. Geometric least square mean (adjusted geometric mean) and adjusted geometric standard error were calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequence', 'period', and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed. Adjusted mean estimates and their difference on log-scale were back-transformed to the original scale.
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Least Squares Mean (Standard Error); unit: nmol*h/L
Arm/Group | BI 1015550 24 mg fed (Test, T) | BI 1015550 24 mg fast (Reference, R)
Number analyzed (Participants) | 11 | 12
nmol*h/L | 4232.24 (NA) — Adjusted geometric standard error = 1.06 | 4131.48 (NA) — Adjusted geometric standard error = 1.06
Statistical Analysis 1: Comparison: BI 1015550 24 mg fed (Test, T) vs BI 1015550 24 mg fast (Reference, R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean (T/R) ratio (%) = 102.44, 90% CI 2-sided [97.80 to 107.30] — To get geometric mean ratio and confidence interval, least square estimates of log-transformed PK endpoint for T and R were back transformed to original scale. Intra-individual geometric coefficient of variance (%) = 5.9

ADVERSE EVENTS:
Time Frame: Adverse events: from drug administration in both periods, up to 168 hours. All-cause mortality: from drug administration until end of study, up to day 15.
Description: Treated set (TS): The treated set included all subjects who were randomised and treated with at least one dose of study drug. The arm "total on treatment" is composed of all the subjects, independently from the treatment received.
Groups:
- BI 1015550 24 mg fed (Test, T): Subjects were treated orally with single dose of BI 1015550 4x6 mg (24 mg) tablets with 240 mL of water under fed condition on day 1.
- BI 1015550 24 mg fast (Reference, R): Subjects were treated orally with single dose of BI 1015550 4x6 mg (24 mg) tablets with 240 mL of water under fasted condition on day 1.
- Total on treatment: Subjects who were treated orally with single dose of BI 1015550 4x6 mg (24 mg) tablets with 240 mL of water under fed / fasted conditions on day 1.
Arm/Group | BI 1015550 24 mg fed (Test, T) | BI 1015550 24 mg fast (Reference, R) | Total on treatment
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/11 | 5/12 | 6/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 1015550 24 mg fed (Test, T) (N=11) | BI 1015550 24 mg fast (Reference, R) (N=12) | Total on treatment (N=12)
Headache (Nervous system disorders) | 1 | 2 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT03302078/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03302078/SAP_001.pdf